CLINICAL TRIAL: NCT04723927
Title: Development of Fall Prediction Model for Older Adults by Analysis of Walking Patterns Based on Multi-faceted Biosignal Data
Brief Title: Development of Fall Prediction Model for Older Adults Based on Multi-faceted Data
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yun-Hee Kim, Principal Investigator, Samsung Medical Center
Other Study IDs: 2020-09-172
Record Dates: First submitted 2021-01-22; First posted 2021-01-26 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Gait
Keywords: Fall prediction model; Gait Pattern; Muscle activity; Brain activity; Cardiopulmonary metabolic cost
MeSH Terms: interventions — Aging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults: The data for motor function and gait pattern analysis was obtained.
  Interventions: Other: Older adults

INTERVENTIONS:
Other: Older adults — The data for motor function and gait pattern analysis was obtained.

SUMMARY:
This study aimed to develop a fall prediction model for older adults by measuring the multi-faceted biosignal data to classify the walking patterns and by identifying causal relationships with the variables that affect the fall.

DETAILED DESCRIPTION:
This study aimed to develop a fall prediction model by measuring the multi-paceted biosignal data for the elderly's physical function and walking to classify the walking patterns of the elderly, and by identifying causal relationships and influences with the variables that affect the fall.

ELIGIBILITY:
Inclusion Criteria:

* Community seniors aged 65 to 84 years
* A person who has no history of central nervous system disease

Exclusion Criteria:

* Older adults who are unable to walk independently due to vision loss, fractures, etc.
* An elderly person who had musculoskeletal history that could cause problems in the function of the lower extremities, such as fractures, within three months before recruitment;
* In case it is difficult to understand the task due to severe cognitive impairment (Korean simplified mental health examination, K-MMSE score 10 or less)
* In the event of a serious mental illness, such as schizophrenia or bipolar disorder;
* In case of severe dizziness and difficulty in pedestrian inspection
* Persons not eligible for examination

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community seniors aged 65 to 84 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Gait analysis | 1 hour
  Gait analysis is a process of measuring and evaluating the walking patterns of patients by using surface electromyograph and motion analysis system.
  All participants perform overground walking to assess the change of kinematic, kinetic and muscle activation using a motion analysis and surface EMG

SECONDARY OUTCOMES:
Change on metabolic energy expenditure | 15 minutes
  All subjects underwent measurements respiratory metabolism energy during treadmill walking at a comfortable speed for 5 minutes.
  It assess the change of metabolic energy expenditure using a portable cardiopulmonary metabolic system (Cosmed K4b², Rome, Italy).
Change on muscle activity | 30 minutes
  All subjects underwent measurements of muscle activity during treadmill walking at a comfortable speed for 5 minutes
Change on brain activity | 30 minutes
  All subjects underwent measurements of brain activity by measuring fNIRS during treadmill walking at a comfortable speed and high speed for 5 minutes
Short Physical Performance Battery (SPPB) | 5 minutes
  The Short Physical Performance Battery (SPPB) is a series of tests used to evaluate lower extremity function and mobility in older people.
Four Square Step Test (FSST) | 5 minutes
  The Four Square Step Test (FSST) is used to assess dynamic stability and the ability of the subject to step over low objects forward, sideways, and backward.
The Timed Up and Go test (TUG) | 5 minutes
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
10 meter walk test (10MWT) | 5 minutes
  Measure of self selected speeds by measuring the time it takes an individual to walk 10 meters. To perform the test, patient walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: "Please walk this distance at your normal pace when I say go."
Modified Bathel index (MBI) | 5 minutes
  The MBI is a measure of activities of daily living, which shows the degree of independence of a patient from any assistance. It covers 10 domains of functioning (activities): bowel control, bladder control, as well as help with grooming, toilet use, feeding, transfers, walking, dressing, climbing stairs, and bathing.
6 minutes walking test (6MWT) | 6 minutes
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
Fall Efficacy Scale (FES) | 5 minutes
  The Falls Efficacy Scale (FES) is a ten-item test rated on a 10-point scale from not confident at all to completely confident.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Chung E, Lee SH, Lee HJ, Kim YH. Comparative study of young-old and old-old people using functional evaluation, gait characteristics, and cardiopulmonary metabolic energy consumption. BMC Geriatr. 2023 Jun 29;23(1):400. doi: 10.1186/s12877-023-04088-6. PMID 37386363